CLINICAL TRIAL: NCT06972719
Title: Patient Centered Education About Hormone Replacement Therapy After Risk Reducing Salpingo-oophorectomy: a Pilot Randomized Controlled Trial
Brief Title: Hormone Replacement Therapy After Risk Reducing Salpingo-oophorectomy
Acronym: BRCA HRT Pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00117007
Record Dates: First submitted 2025-04-30; First posted 2025-05-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-08

CONDITIONS: BRCA1 Mutation; BRCA2 Mutation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Placebo Comparator): The control arm will receive standard counseling regarding post operative HRT by their gynecologic oncologist during their visit, as well as standardized written education in their after-visit summary.
  Interventions: Behavioral: SOC Arm
- Experimental (Experimental): The experimental arm will receive standard verbal counseling and written education plus the video-based educational aid describing the risks and benefits of HRT.
  Interventions: Behavioral: Experimental Arm

INTERVENTIONS:
Behavioral: Experimental Arm — Participants will be randomized to SOC plus the video.
  Arms: Experimental
Behavioral: SOC Arm — Participants will be randomized to SOC counseling.
  Arms: Standard of Care

SUMMARY:
The goal of this study is to develop an educational aid about hormone replacement therapy that physicians can share with patients as part of their pre-surgical counseling for a risk-reducing salpingo-oophorectomy (RRSO).

DETAILED DESCRIPTION:
The proposed randomized study seeks to enroll 50 individuals from gynecologic oncology and high-risk breast clinics who are actively planning RRSO. Participants will be randomized to usual provider education versus usual education plus video education. The researchers will assess participants' level of conflict around the decision to use HRT, their satisfaction with their decision, their satisfaction with their counseling, and their postoperative decision regarding HRT. This project will provide pilot data for a larger randomized trial. Ultimately, the investigators seek to create a comprehensive aid for education and values clarification, with the aim of improving informed decision making for individuals with BRCA1-2 mutations.

ELIGIBILITY:
Inclusion Criteria:

* BRCA1 or BRCA2 germline mutation
* scheduled for a risk-reducing salpingo-oophorectomy (RRSO) by Duke Gynecologic Oncologist
* premenopausal

Exclusion Criteria:

* personal history of cancer
* postmenopausal
* >50 years old
* unable to provide informed consent in English

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Decisional Conflict pre-randomization | Baseline, pre-randomization
  The Decisional Conflict Scale ranges from 16 to 80 with a higher score indicating greater conflict with the decision.
Decisional Conflict post-intervention | Immediately after the intervention
  Decisional conflict will be reassessed preoperatively after all materials have been reviewed. The Decisional Conflict Scale ranges from 16 to 80 with a higher score indicating greater conflict with the decision.
Decisional Conflict post-operatively | 2-6 weeks post op
  Decisional conflict will be reassessed postoperatively. The Decisional Conflict Scale ranges from 16 to 80 with a higher score indicating greater conflict with the decision.
Satisfaction with Counseling | 2-6 weeks post op
  a Likert-scale questionnaire to assess their satisfaction with their preoperative counseling.
Satisfaction with Decision | 3-6 months post op
  The Satisfaction with Decision scale ranges from 6 to 30 with higher scores indicating greater satisfaction with their decision.

SECONDARY OUTCOMES:
Number of participants who decide to take HRT | 3-6 months post op
  Number of participants who decide to take HRT
Number of participants who decide to take estrogen, a progesterone, or an estrogen + progesterone medication | 3-6 months post op
  Number of participants who decide to take estrogen, a progesterone, or an estrogen + progesterone medication

CONTACTS AND LOCATIONS:
Overall Officials: Laura Havrilesky, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No